CLINICAL TRIAL: NCT01069380
Title: Resting Metabolic Rate in Chronic Bed-Ridden Patients
Acronym: RMR
Status: Terminated | Type: Observational
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Reuth Research Institute, Research coordinator, Reuth Rehabilitation Hospital
Other Study IDs: RMC2010-4CTIL
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Chronic Disease
Keywords: resting metabolic rate; bed ridden, vegetative; low conscious; minimal conscious state; immobilized; resting energy expenditure
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Research objective: to measure resting metabolic rate (REE) in long term, bed ridden, chronically ill patients and to compare their measured energy needs to standard REE equations

DETAILED DESCRIPTION:
Are standard REE equations suitable for estimating resting metabolic rate in long term, bed ridden, chronically ill patients?

Research objective: to measure resting metabolic rate (REE) in long term, bed ridden, chronically ill patients and to compare their measured energy needs to standard REE equations

ELIGIBILITY:
Inclusion Criteria:

* Age (years): 18-30, 31-60, 61-74, 75-100
* Confinement to bed at least for a year

Exclusion Criteria:

* Mechanical ventilation
* Tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronically bed ridden patients for at least 1 year, hospitaqlized in REUTH MEDICAL CENTER
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09-10 (Actual); Study Completion 2011-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham AL Lazary, MD, Principal Investigator — Reuth Rehabilitation Hospital
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel